CLINICAL TRIAL: NCT00455117
Title: Phase Four Study of Intravenous Parecoxib on Post-craniotomy Pain
Brief Title: Effect of Parecoxib on Post-craniotomy Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Parecoxib_HREC2006.133
Record Dates: First submitted 2007-04-01; First posted 2007-04-03 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Anaesthesia
Keywords: analgesia; pain; neurosurgery; NSAIDS; parecoxib; morphine consumption
MeSH Terms: conditions — Agnosia; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo (2 ml normal saline) administered intravenously at dural closure during craniotomy
  Interventions: Drug: Intravenous Parecoxib ('Dynastat' Pfizer)
- 2 (Active Comparator): parecoxib 40 mg in 2 ml normal saline administered intravenously at dural closure during craniotomy
  Interventions: Drug: Intravenous Parecoxib ('Dynastat' Pfizer)

INTERVENTIONS:
Drug: Intravenous Parecoxib ('Dynastat' Pfizer) — parecoxib or placebo
  Other Names: Intravenous parecoxib ("Dynastat" Pfizer)

SUMMARY:
Aim of this trial:

To investigate whether post-craniotomy analgesia with (i) intravenous (IV) parecoxib plus intravenous paracetamol is superior to (ii) intravenous paracetamol alone.

Study Hypothesis:

Post-operative analgesia with intravenous parecoxib in combination with intravenous paracetamol will be superior to intravenous paracetamol alone.

DETAILED DESCRIPTION:
Neurosurgical patients undergoing brain procedures (craniotomy patients) are known to suffer moderately severe postoperative pain and high rates of post-operative nausea and vomiting. Post-craniotomy pain is poorly treated with more than 50% of craniotomy patients experiencing postoperative pain of moderate or severe intensity. Fear of drug complications such as sedation, respiratory depression, seizures and intracranial bleeding has inhibited prescribing of effective pain treatment.Non-steroidal anti-inflammatory drugs (NSAIDS) are known to be effective analgesics in the peri-operative period however there use in cranial neurosurgery has been limited due to risk of bleeding. Parecoxib is an injectable form of NSAID that works through inhibiting cyclo-oxygenase type-2 (COX-2). The main benefit of COX-2 inhibitors is that they have minimal inhibition of platelet function and therefore minimal risk of increased bleeding.This project aims to evaluate whether parecoxib is an effective pain reliever (analgesic) after brain surgery. Patients aged 18-65 years presenting for elective craniotomy will be randomly allocated to two different analgesic programs (i) IV parecoxib and IV paracetamol or (ii) IV paracetamol. All patients will receive a standardised anaesthetic. Scalp infiltration, using 20mls of local anesthetic (bupivacaine 0.5% with adrenaline), will occur prior to skin incision. Intermittent morphine administration will used post-operatively to ensure adequate analgesia in each arm of the trial. Immediate post-operative adjunctive analgesia will be provided with nurse administered IV morphine in the post-anaesthetic care unit (PACU) as per protocol (RMH protocol for opioid titration), followed by patient controlled analgesia (PCA) morphine once the verbal rating scale is < 4 (rating out of ten). A score of less than four is considered to be mild pain. PCA will be continued for the first twenty-four hours then discontinued. Patients will then receive strict oral paracetamol and nurse administered IV morphine as required. The primary study endpoint will be morphine consumption in the first 24 hours. Data will be analysed on an intention to treat basis. Continuous variables will be graphed to determine their distribution. Normally distributed variables will be described using mean and standard deviation and compared using Student's t-tests. Skewed variables will be described using median and range (or interquartile range) and compared using Wilcoxon rank sum tests. A p-value les than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Supratentorial craniotomy, glasgow coma scale 15

Exclusion Criteria:

* Chronic pain,
* Chronic opioid use.
* History of significant alcohol or benzodiazepine (BZD) use,
* Inability to speak English,
* Pre-operative aphasia or dysphasia,
* Renal impairment (Creatinine level > 0.1),
* Asthma (or evidence of reversible airway obstruction,
* Known ischaemic heart disease or cerebrovascular disease,
* American Society of Anaesthesiologists (ASA) grade IV or V,
* Allergy to any study drug (paracetamol, parecoxib, sulphas, morphine, bupivacaine, propofol, remifentanil;
* Administration of oral paracetamol within previous 8 hours.
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Morphine consumption in 24 hour period. | 24 hours after surgery

SECONDARY OUTCOMES:
Immediate post-operative hypertension (first 2 hours) | 24 hours after surgery
Pain scores at zero (time of extubation), 1, 2, 4, 12, 24 hours post operatively | 24 hours after surgery
Analgesic efficacy at 24 hours | 24 hours after surgery
Incidence of post-operative nausea and vomiting (first 24 hours) | 24 hours after surgery
Sedation or respiratory depression (first 24 hours) | 24 hours after surgery
Safety Monitoring (Serious adverse side effects) | 24 hours after surgery
Post-operative AMI | 24 hours after surgery
Post-operative renal failure | 24 hours after surgery
Post-operative thromboembolic stroke | 24 hours after surgery
Post-operative intracranial haemorrhage | 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daryl L Williams, MBBS, Principal Investigator — Director of Anaesthesia, Royal Melbourne Hospital
Locations (1):
- Royal Melbourne Hospital, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Williams DL, Pemberton E, Leslie K. Effect of intravenous parecoxib on post-craniotomy pain. Br J Anaesth. 2011 Sep;107(3):398-403. doi: 10.1093/bja/aer223. PMID 21841050